## **IRB-Approved Consent Forms for:**

Development and Pilot Trial of an Intervention to Reduce Disclosure Recipients Negative Social Reactions and Victims Psychological Distress and Problem Drinking

NCT03488927

Last approved April 1st, 2019

## **Contents:**

Informed consent: Initial survey
Informed consent: Program
Informed consent: Post-test survey
Informed consent: victim

## **Informed Consent: Initial survey**

## IRB #6745E

#### **Fast Facts**

- ✓ You are invited to take a few surveys and to participate in an educational workshop!
- ✓ Participation in the project is voluntary and optional.
- ✓ Your answers are confidential, with some exceptions (listed below). You will receive \$15 gift card for participating in the online survey today, \$25 for participating in an in-person survey after the first 90-minute workshop, \$25 for participating in an in-person survey after the second 60-minute workshop, and \$25 for participating in the final online survey. You can skip questions and still get the monetary incentive. You can earn up to \$100 in total.
- ✓ If you complete all parts of the study, you will be entered to win one of two \$500 Visa gift cards!!
- ✓ By agreeing to participate today, you are agreeing to participate in all four components of the study, although you may withdraw at any time.
- ✓ Read BELOW for the full details to decide if you are willing to participate!

In the details below, we will mostly focus on today's survey. At each phase of the research, we will provide more detail about that phase.

**Purpose:** The purpose of this project is to examine what college students think about a curriculum titled *Supporting Survivors and Self: An Educational Curriculum for Social Supports of Survivors of Partner Abuse and Sexual Aggression.* If you choose to participate you will be asked to complete an online survey and another survey in six months. You will also be asked to participate two educational workshops. You might also be asked to do a combination of the following: participate in a one-on-one interview and/or tell friends/peers you have helped to get in touch with us about participating in this project. All of these activities are voluntary and optional. You will receive monetary compensation for your participation in each part of the project. The ultimate goal of this project is to see how this program is working and to make it better so that it is useful to college students. We are hoping to recruit approximately 1000 people to participate in this project, and a minimum of 700 people. **You must be an undergraduate at UNH student between the ages of 18 to 24 to participate. DO NOT FORWARD THE INVITATION OR SHARE THE SURVEY LINK WITH OTHER STUDENTS.** 

**Description of the Study:** If you decide to be part of this initial survey, you will be asked to:

- 1. Complete an online survey that will take about 20 minutes; the survey will ask you things about yourself, like demographics, your attitudes, and also about unwanted sexual, physical, and emotional experiences that you have had or that your friends/peers have had.
- 2. Provide us with your contact information so that we can send you gift card information and find a time for you to complete the educational workshops.
- 3. Please only complete the initial survey if you are also planning to attend the workshops.

**Voluntary Participation and Right to Withdraw:** Being in this study is voluntary, which means you don't have to be in the study. If you start the study, you can drop out at any time. You can stop answering questions during the survey. You must get to the end of the survey in order to get the \$15 gift card. You can skip questions and still get the \$15; you just need to get to the end of the survey.

## **Confidentiality:**

- (1) The researcher plans to keep what you say and answer confidential. This means they will keep your answers private and not share them with anyone else. You will not write your name on the survey.
- (2) When the researchers go to tell other researchers what they found they will talk about what groups of students said or will talk about words students said without using their names. We will never share information that might identify a student in publications or presentations.
- (3) However, there are some exceptions to confidentiality, which we outline below. It is important that you know that NONE of the questions we will ask you in the survey today (or in future surveys or interviews) will ask you to tell us about this level of detail and so we urge you not to write any of the things listed below in open response questions (e.g., contact information) on the survey or tell us by email, phone, or in person. If you want to make the university aware of any such issues so that they can take action, please consult with the UNH TIX Coordinator, UNH police, and any other trusted UNH official. If you would like confidential support to help manage these issues but don't want the university to be notified or to take action, please contact UNH Psychological and Counseling Services, UNH Health and Wellness, or the UNH Sexual Harassment and Rape Prevention Program (SHARPP).
  - If you tell us that you are thinking about or plan to seriously hurt or kill yourself or someone else, we will notify the UNH behavioral intervention team and/or the UNH police.
  - If you tell us about a child (a person currently under 18) or elder who is being abused or a
    person who is abusing a child or elder, we will notify the NH Department of Health and
    Human Services. Child and elder abuse include words or actions that cause harm, potential
    harm, or threat of harm to a child or elder, including physical, sexual, and psychological
    abuse.
  - If you tell us about student hazing, we will notify the UNH police. Hazing is defined by UNH as: "an act directed toward a student, or any coercion or intimidation of a student to act or to participate in an act, for the purpose of initiation or admission into, affiliation with, or as a condition for continued membership in, a group or organization, when (1) such act is likely or would be perceived by a reasonable person as likely to cause physical or psychological injury to any person; or (2) destroys or removes public or private property."
  - If you tell us about a student being sexually harassed or sexually assaulted by a USNH employee, we will notify University Police and the Title IX Coordinator (Director of the Affirmative Action and Equity Office).
- (4) Please note that confidentiality of disclosures of sexual violence and sexual harassment made in this research project extends only to the research work, and not to outside discussions with the researchers.
- (5) Also, the University of New Hampshire Institutional Review Board can see the data in some cases. An example would be if you complained to the University that you did not like something about the survey or research study. Because none of the data we get from you will have your name, the University cannot see your answers but might decide to look at all of the answers participants gave us without knowing their names.

- (6) All of your answers from the surveys will be stored as a number, not with your name. All test surveys, notes, and records from this project will be kept in a locked room in either a locked cabinet or on a secured network in Dr. Edwards' research lab at the University of New Hampshire.
- (7) This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see above); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects. The Certificate of Confidentiality will not be used to prevent disclosure as required by federal, state, or local law in cases of: threats of serious injury to self or others, child or elder abuse, hazing, or sexual violence perpetrated by a UNSH employee. The Certificate cannot be used to refuse a request for information from personnel from the agency sponsoring the project that is needed for auditing or program evaluation by the National Institutes of Health, which is funding this project. You should understand that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to any other person not connected with the research, you must provide consent to allow the researchers to release it.
- (8) Please note that if you win the drawing and accept the \$500 gift card, you will be asked to provide some personal information to receive the card; this information depends on resident status. Please contact UNH's Academic Affairs Business Service Center for more details.

**Potential Benefits:** A lot of college students say that they enjoy participating in research because they learn about themselves and feel proud to be part of science that helps others. The information you provide will also help us to create programs for college students.

**Potential Risks:** Because you will be asked to think about things like dating and sexual relationships, including unwanted experiences, you might feel sad or shy or scared talking about these things. However, most students do not report being upset by these types of questions. For students who do report being upset, usually they only report being a little upset and for just a little bit of time. Remember that you do not have to answer any questions you do not want to answer. We will provide you with a PDF document that has information about counseling and support services that are available to students. Other risks, such as needing to break confidentiality, were reviewed above. Finally, any communication via the Internet poses minimal risk of a breach of confidentiality.

**Future Questions and Concerns:** The University of New Hampshire's Institutional Review Board for the Protection of Human Subjects in Research has approved the use of human subjects in this study. If you have any questions about this research project or would like more information before, during, or after

| the study, you may contact Dr. Katie Edwards by phone (603-862-3720) or email |
|---|
| (Katie.Edwards@unh.edu). If you have questions about your rights as a research subject, you may |
| contact Melissa McGee in UNH Research Integrity Services at 603-862-2005 or Melissa.McGee@unh.edu |
| to discuss them. |

| Please click one of the options below: |
|----------------------------------------|
| Yes, I agree to take the survey. |
| No, I do not want to take the survey |

## **Informed Consent: Program**

## IRB #6745E

#### **Fast Facts**

- ✓ You are invited to participate in an educational workshop!
- ✓ We will NEVER ask you to disclose violence victimization. If you do disclose violence victimization, we are mandated reporters in some situations not others; please read below for more details.
- ✓ You will receive \$25 cash after the session.
- ✓ Read below for the full details to decide if you are willing to participate!

**Purpose:** The purpose of this project is to examine what college students think about a curriculum titled *Supporting Survivors and Self: An Educational Curriculum for Social Supports of Survivors of Partner Abuse and Sexual Aggression.* You will be asked to complete two sessions of an educational program. After each of the two sessions you will be asked to fill out surveys to tell us what you think about the program. You will also be asked to complete an online survey about six months later. The ultimate goal of this project is to see how this program is working and to make it better so that it is useful to college students. We are hoping to recruit approximately 1000 people to participate in this project, and a minimum of 700 people. **You must be and undergraduate student between the ages of 18 to 24 to participate.** 

**Description of the Study:** If you decide to be part of this initial survey, you will be asked to:

- 1. Participate in an educational program that will talk to you about how to help friends with upsetting sexual and relationship experiences, and will involve group discussions. The educational program will be audio-recorded; the reason we will record the sessions is so that the researchers can review the sessions to make the program better and give feedback to the people teaching the program. Please note that these sessions will include facilitators and participants of all genders.
- 2. Fill out surveys after each of the two sessions telling us what you think about the program; you will be paid \$25 for each of the two surveys that you complete. You cannot fill out these surveys if you do not come to the program sessions.
- 3. Please note that you must be on time to the workshop to participate. Once we have collected signed consent forms, we cannot allow any more participants to enter the workshop, because they have consented.

We might ask you to share information with your friends about the project. We might also ask you to participate in a one on one conversation with us about the program. All of this, like all parts of the study are voluntary, meaning you can say no.

**Voluntary Participation and Right to Withdraw:** Being in this study is voluntary, which means you don't have to be in the study. If you start the study, you can drop out at any time. You can stop answering questions during the survey. You must get to the end of each of the study sessions in order to get the \$25. You can skip questions and still get the \$25.

## **Confidentiality:**

- (1) The researcher plans to keep what you say and answer confidential. This means they will keep your answers private and not share them with anyone else. You will not write your name on the survey. We will not record names when we transcribe the audio-recorded group discussion.
- (2) When the researchers go to tell other researchers what they found they will talk about what groups of students said or will talk about words or quotes students said without using their names. We will never share information that might identify a student in publications or presentations.
- (3) However, there are some exceptions to confidentiality, which we outline below. It is important that you know that NONE of the questions we will ask you in any of the surveys or in questions posed in the group discussion will ask you to tell us about this level of detail and so we urge you not to make disclosures about the below in the research survey. If you want to make the university aware of any such issues so that they can take action, please consult with the UNH TIX Coordinator, UNH police, and any other trusted UNH official. If you would like confidential support to help manage these issues but don't want the university to be notified or to take action, please contact UNH Psychological and Counseling Services, UNH Health and Wellness, or the UNH Sexual Harassment and Rape Prevention Program (SHARPP).
  - a. If you tell us that you are thinking about or plan to seriously hurt or kill yourself or someone else, we will notify the UNH behavioral intervention team and/or the UNH police.
  - b. If you tell us about a child (a person currently under 18) or elder who is being abused or a person who is abusing a child or elder, we will notify the NH Department of Health and Human Services. Child and elder abuse include words or actions that cause harm, potential harm, or threat of harm to a child or elder, including physical, sexual, and psychological abuse.
  - c. If you tell us about student hazing, we will notify the UNH police. Hazing is defined by UNH as: "an act directed toward a student, or any coercion or intimidation of a student to act or to participate in an act, for the purpose of initiation or admission into, affiliation with, or as a condition for continued membership in, a group or organization, when (1) such act is likely or would be perceived by a reasonable person as likely to cause physical or psychological injury to any person; or (2) destroys or removes public or private property."
  - d. If you tell us about a student being sexually harassed or sexually assaulted by a UNH faculty or staff member, we will notify University Police or the Title IX Coordinator (Director of the Affirmative Action and Equity Office).
- (4) <u>Please note that confidentiality of disclosures of sexual violence and sexual harassment made in this research project extends only to the research work, and not to outside discussions with the researchers.</u>
- (5) Note to Student Workers: Although you may normally be required to report to the UNH Title IX Coordinator and UNH Police any disclosures made to you by other students about sexual violence and/or sexual harassment because of your UNH job (e.g., Resident Assistants, Teaching Assistants), you are NOT required to make such reports based upon any disclosures made by other students that come to your attention because of your participation in any group discussion activities associated with this research project. You should not solicit participation in this project by any individual who you know through your job.
- (6) Also, the University of New Hampshire Institutional Review Board can see the data in some cases. An example would be if you complained to the University that you did not like something about the

- survey or research study. Because none of the data we get from you will have your name, the University cannot see your answers but might decide to look at all of the answers participants gave us without knowing their names.
- (7) All of your answers from the surveys will be stored as a number, not with your name. All test surveys, notes, and records from this project will be kept in a locked room in either a locked cabinet or on a secured network in Dr. Edwards' research lab at the University of New Hampshire.
- (8) This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see above); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects. The Certificate of Confidentiality will not be used to prevent disclosure as required by federal, state, or local law in cases of: threats of serious injury to self or others, child or elder abuse, hazing, or sexual violence perpetrated by a UNSH employee. The Certificate cannot be used to refuse a request for information from personnel from the agency sponsoring the project, that is needed for auditing or program evaluation by the National Institutes of Health, which is funding this project. You should understand that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to any other person not connected with the research, you must provide consent to allow the researchers to release it.

**Potential Benefits:** A lot of college students say that they enjoy participating in research because they learn about themselves and feel proud to be part of science that helps others. The information you provide will also help us to create programs for college students.

**Potential Risks:** Because you will be asked to think about things like dating and sexual relationships, you might feel sad or shy or scared talking about these things. However, most students do not report being upset by these types of questions. For students who do report being upset, usually they only report being a little upset and for just a little bit of time. Remember that you do not have to answer any questions you do not want to answer. Participation in the group discussion and program is voluntary. We will give you a sheet of paper that has information about counseling and support services that are available to students. Other risks such as needing to break confidentiality was reviewed above. Finally, any communication via the Internet poses minimal risk of a breach of confidentiality.

**Future Questions and Concerns:** The University of New Hampshire's Institutional Review Board for the Protection of Human Subjects in Research has approved the use of human subjects in this study. If you have any questions about this research project or would like more information before, during, or after the study, you may contact Dr. Katie Edwards by phone (603-862-3720) or email (Katie.Edwards@unh.edu). If you have questions about your rights as a research subject, you may

contact Melissa McGee in UNH Research Integrity Services at 603-862-2005 or Melissa.McGee@unh.edu to discuss them.

# **CONSENT TO PARTICIPATE**

| I,participate in this research | (print name) CONSENT/AGREE to project |
|---|---|
| Participant's Signature | <br>Date |
| CONFIDENTIALITY PROMI | SE |
| | (print name) AGREE to keep today's eaning that I will not tell other people what ring the discussion. |
| Participant's Signature | <br> |

## **Informed Consent: Post-test survey**

## IRB #6745E

- ✓ You are invited to take a survey just like the one you took about six months ago!
- ✓ The purpose of this project is to examine what college students think about a curriculum titled Supporting Survivors and Self: An Educational Curriculum for Social Supports of Survivors of Partner Abuse and Sexual Aggression.
- ✓ Participation in this project is voluntary and optional.

No, I do not want to take the survey

- ✓ Please do not forward this invitation or share the survey link with other students.
- ✓ You will receive \$25 gift card for finishing the survey. You can skip questions and still get the \$25, but you have to make it to the end of the survey.
- ✓ In addition to the survey, you might also be asked to, if you want to, tell friends/peers you have helped to get in touch with us about participating in this project. If so, we will ask you to reach out to friends to participate in the study for one additional gift card incentive (\$10). We will call you to offer guidance on how to invite friends. This part, like all parts of the research, are voluntary. If you choose to participate in this part, we will ask you to report back to us, via a short survey, how many people you told. We will then send you the additional gift card.
- ✓ Your answers are confidential, with the same exceptions as we listed in the first survey (harm to self/or others, child abuse, elder abuse, hazing, and sexual harassment or assault perpetrated by a USNH employee).
- ✓ We will provide you with a PDF document that has information about counseling and support services that are available to students.
- ✓ The University of New Hampshire's Institutional Review Board for the Protection of Human Subjects in Research has approved the use of human subjects in this study. If you have any questions about this research project or would like more information before, during, or after the study, you may contact Dr. Katie Edwards by phone (603-862-3720) or email (<a href="Katie.Edwards@unh.edu">Katie.Edwards@unh.edu</a>). If you have questions about your rights as a research subject, you may contact Melissa McGee in UNH Research Integrity Services at 603-862-2005 or Melissa.McGee@unh.edu to discuss them.

| Please click one of the options below: |
|----------------------------------------|
| Yes, I agree to take the survey. |

## **Informed Consent: Victim survey**

#### IRB #6745E

Purpose: The purpose of this project is to examine how friends support friends who tell them about unwanted sexual and relationship experiences. We anticipate a minimum of 20 other individuals will take this survey (although we are aiming for about 100 individuals). You must be over the age of 18 to participate. DO NOT FORWARD THE INVITATION OR SHARE THE SURVEY LINK WITH OTHER STUDENTS.

Description of the Study: If you decide to be part of this survey, you will be asked to: Complete an online survey about how other people responded to your unwanted experiences, how you are feeling including psychological symptoms, some details about negative sexual and relationship experiences, and about substance use. You are required to answer these questions in this survey, to allow us to accurately analyze the impact of the program on students such as yourself. If you are not comfortable with answering these types of questions, you should not consent to move forward with the survey. Also, the link you have been given is connected to the name of the person who told you about this survey, but only so that we can confirm that the link was sent by someone who participated in the initial phase of the project. We will destroy our list of those participants once all the data is collected. If you have questions, please contact the research team at sss.research@unh.edu or at 603-285-8237.

At the beginning of the survey, you will be asked several screening questions. If there questions indicate you are eligible, you can move forward to through the survey and then receive the incentive. If these questions indicate you are not eligible, you will not be able to take the survey, and thus, will not receive the incentive. Please note that if you have also taken the other SSS survey that asks about your reactions to disclosure, you cannot also get a gift card for taking this survey.

Voluntary Participation and Right to Withdraw: Being in this study is voluntary, which means you don't have to be in the study. If you start the study, you can drop out at any time. You can stop answering questions during the survey. You must get to the end of the survey in order to get the \$25.

Confidentiality: (1) The researcher plans to keep what you say and answers confidential. This means they will keep your answers private and not share them with anyone else. You will not write your name on the survey. (2) When the researchers go to tell other researchers what they found they will talk about what groups of students said or will talk about words students said without using their names. We will never share information that might identify a student in publications or presentations.

(3) However, there are some exceptions to confidentiality, which we outline below. It is important that you know that NONE of the questions we will ask you in the survey today will ask you to tell us about this level of detail and so we urge you not to write any of the things listed below in open response questions (e.g., contact information) on the survey or tell us by email, phone, or in person. If you want to make the university aware of any such issues so that they can take action, please consult with the UNH Title IX Coordinator, UNH police, and any other trusted UNH official. If you would like confidential support to help manage these issues but don't want the university to be notified or to take action, please contact UNH Psychological and Counseling Services, UNH Health and Wellness, or the UNH Sexual Harassment and Rape Prevention Program (SHARPP). Links to this information will be available after the survey. a. If you tell us that you are thinking about or plan to seriously hurt or kill yourself or someone else, we will notify the UNH behavioral intervention team and/or the UNH police. b. If you

tell us about a child (a person currently under 18) or elder who is being abused or a person who is abusing a child or elder, we will notify the NH Department of Health and Human Services. Child and elder abuse include words or actions that cause harm, potential harm, or threat of harm to a child or elder, including physical, sexual, and psychological abuse. c. If you tell us about student hazing, we will notify the UNH police. Hazing is defined by UNH as: "an act directed toward a student, or any coercion or intimidation of a student to act or to participate in an act, for the purpose of initiation or admission into, affiliation with, or as a condition for continued membership in, a group or organization, when (1) such act is likely or would be perceived by a reasonable person as likely to cause physical or psychological injury to any person; or (2) destroys or removes public or private property." d. tell us about a student being sexually harassed or sexually assaulted by a USNH employee, we will notify University Police and the Title IX Coordinator (Director of the Affirmative Action and Equity Office). (4) Please note that confidentiality of disclosures of sexual violence and dating violence made in this research project extends only to the research work, and not to outside discussions with the researchers. (5) Also, the University of New Hampshire Institutional Review Board can see the data in some cases. An example would be if you complained to the University that you did not like something about the survey or research study. Because none of the data we get from you will have your name, the University cannot see your answers but might decide to look at all of the answers participants gave us without knowing their names. (6) All of your answers from the surveys will be stored as a number, not with your name. All test surveys, notes, and records from this project will be kept in a locked room in either a locked cabinet or on a secured network in Dr. Edwards' research lab at the University of New Hampshire. (7) This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see above); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects. The Certificate of Confidentiality will not be used to prevent disclosure as required by federal, state, or local law in cases of: threats of serious injury to self or others, child or elder abuse, hazing, or sexual violence perpetrated by a USNH employee. The Certificate cannot be

used to refuse a request for information from personnel from the agency sponsoring the project that is needed for auditing or program evaluation by the National Institutes of Health, which is funding this project. You should understand that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to any other person not connected with the research, you must provide consent to allow the researchers to release it.

Potential Benefits: A lot of college students say that they enjoy participating in research because they learn about themselves and appreciate the opportunity to contribute to science. The information you provide will also help us to create programs for college students.

Potential Risks: Because you will be asked to think about things like negative dating and sexual relationship expereinces, you might feel upset, reluctant or anxious about these things. However, most students do not report being upset by these types of questions. For participants who do report being upset, usually they only report being a little upset and for just a little bit of time. Remember that you do not have to answer any questions you do not want to answer. We will provide you with a PDF document that has information about counseling and support services that are available to students. Other risks such as needing to break confidentiality was reviewed above. Finally, any communication via the Internet poses minimal risk of a breach of confidentiality.

Future Questions and Concerns: The University of New Hampshire's Institutional Review Board for the Protection of Human Subjects in Research has approved the use of human subjects in this study. If you have any questions about this research project or would like more information before, during, or after the study, you may contact Dr. Katie Edwards by phone (603-862-3720) or email (Katie.Edwards@unh.edu). If you have questions about your rights as a research subject, you may contact Melissa McGee in UNH Research Integrity Services at 603-862-2005 or Melissa.McGee@unh.edu to discuss them.

Vic\_Consent4. Please click one of the options below:

If you are not sure yet and have questions, please contact the SSS team at SSS.research@unh.edu or at 603.285.8237 before answering this question.